CLINICAL TRIAL: NCT02045407
Title: Computed Tomography Angiography Accuracy in Brain Death Diagnosis
Status: Completed | Type: Observational
Sponsor: Sergio Brasil, MD MSc (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Sergio Brasil, MD MSc, MD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: 12500913400000068
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Brain Death
Keywords: Brain Death; Neurological Death; Cerebral circulatory arrest; Computed Tomography Angiography
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the reliability of computed tomography angiography (CTA) to diagnose brain death, face of several conditions that make impossible to define such diagnosis using clinical criteria exclusively.

DETAILED DESCRIPTION:
Critically ill patients, presenting Glasgow Coma Score 5 or lower, will be submitted to the Computed Tomography Angiography (CTA) of the skull assessment, and follow a clinical evaluation for brain death, additionally, transcranial Doppler would be applied as the gold standard for brain death.

We will exclude patients whose do not can be submitted to contrast injection, or if a brain death clinical evaluation has been performed prior the CTA.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any age or sex with brain death suspicion raised, before clinical test.
* Comatose patients presenting Glasgow Coma Score as or under 5 points, under sedative agents or not.

Exclusion Criteria:

* Brain dead patients clinically confirmed.
* Contraindications to the use of contrast medium (renal failure or allergy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any genre or age.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Assess the presence or absence of contrast medium filling of the intracranial vessels in comatose patients. | 1 year
  After excluding confounding factors, we will submit comatose patients to CTA. Immediately after the exam, we will perform clinical evaluation for brain death and calculate CTA sensibility and specificity for this diagnosis. Time between these two interventions will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Brasil, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP., São Paulo, Brazil

REFERENCES:
- [Result] Welschehold S, Kerz T, Boor S, Reuland K, Thomke F, Reuland A, Beyer C, Tschan C, Wagner W, Muller-Forell W, Giese A. Computed tomographic angiography as a useful adjunct in the diagnosis of brain death. J Trauma Acute Care Surg. 2013 May;74(5):1279-85. doi: 10.1097/TA.0b013e31828c46ba. PMID 23609279
- [Result] Welschehold S, Kerz T, Boor S, Reuland K, Thomke F, Reuland A, Beyer C, Wagner W, Muller-Forell W, Giese A. Detection of intracranial circulatory arrest in brain death using cranial CT-angiography. Eur J Neurol. 2013 Jan;20(1):173-9. doi: 10.1111/j.1468-1331.2012.03826.x. Epub 2012 Jul 12. PMID 22788547
- [Result] Rieke A, Regli B, Mattle HP, Brekenfeld C, Gralla J, Schroth G, Ozdoba C. Computed tomography angiography (CTA) to prove circulatory arrest for the diagnosis of brain death in the context of organ transplantation. Swiss Med Wkly. 2011 Oct 4;141:w13261. doi: 10.4414/smw.2011.13261. eCollection 2011. PMID 21971739
- [Result] Bohatyrewicz R, Sawicki M, Walecka A, Walecki J, Rowinski O, Bohatyrewicz A, Kanski A, Czajkowski Z, Krzysztalowski A, Solek-Pastuszka J, Zukowski M, Marzec-Lewenstein E, Wojtaszek M. Computed tomographic angiography and perfusion in the diagnosis of brain death. Transplant Proc. 2010 Dec;42(10):3941-6. doi: 10.1016/j.transproceed.2010.09.143. PMID 21168593
- [Result] Berenguer CM, Davis FE, Howington JU. Brain death confirmation: comparison of computed tomographic angiography with nuclear medicine perfusion scan. J Trauma. 2010 Mar;68(3):553-9. doi: 10.1097/TA.0b013e3181cef18a. PMID 20220416
- [Result] Escudero D, Otero J, Marques L, Parra D, Gonzalo JA, Albaiceta GM, Cofino L, Blanco A, Vega P, Murias E, Meilan A, Roger RL, Taboada F. Diagnosing brain death by CT perfusion and multislice CT angiography. Neurocrit Care. 2009;11(2):261-71. doi: 10.1007/s12028-009-9243-7. Epub 2009 Jun 30. PMID 19565357
- [Result] Frampas E, Videcoq M, de Kerviler E, Ricolfi F, Kuoch V, Mourey F, Tenaillon A, Dupas B. CT angiography for brain death diagnosis. AJNR Am J Neuroradiol. 2009 Sep;30(8):1566-70. doi: 10.3174/ajnr.A1614. Epub 2009 Apr 30. PMID 19406767
- [Result] Dupas B, Gayet-Delacroix M, Villers D, Antonioli D, Veccherini MF, Soulillou JP. Diagnosis of brain death using two-phase spiral CT. AJNR Am J Neuroradiol. 1998 Apr;19(4):641-7. PMID 9576648
- [Result] Leclerc X, Taschner CA, Vidal A, Strecker G, Savage J, Gauvrit JY, Pruvo JP. The role of spiral CT for the assessment of the intracranial circulation in suspected brain-death. J Neuroradiol. 2006 Apr;33(2):90-5. doi: 10.1016/s0150-9861(06)77237-6. PMID 16733422
- [Result] Combes JC, Chomel A, Ricolfi F, d'Athis P, Freysz M. Reliability of computed tomographic angiography in the diagnosis of brain death. Transplant Proc. 2007 Jan-Feb;39(1):16-20. doi: 10.1016/j.transproceed.2006.10.204. PMID 17275466
- [Result] Quesnel C, Fulgencio JP, Adrie C, Marro B, Payen L, Lembert N, El Metaoua S, Bonnet F. Limitations of computed tomographic angiography in the diagnosis of brain death. Intensive Care Med. 2007 Dec;33(12):2129-35. doi: 10.1007/s00134-007-0789-6. Epub 2007 Jul 21. PMID 17643226